CLINICAL TRIAL: NCT02567799
Title: A Phase I/II Clinical Study Evaluating the Safety and Effectiveness of BIO 300 Oral Suspension in Patients Receiving Chemoradiation Therapy for Non-Small Cell Lung Cancer (NSCLC)
Brief Title: BIO 300 Non-Small Cell Lung Cancer Study
Acronym: NSCLC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Humanetics Corporation (Industry)
Collaborators: National Cancer Institute (NCI) (NIH); Henry Ford Health System (Other); Medical College of Wisconsin (Other); University of Maryland, Baltimore (Other); Milwaukee VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CL0101-01; HHSN261201200078C (Other Grant/Funding Number: NCI)
Record Dates: First submitted 2015-07-09; First posted 2015-10-05 (Estimated); Results first posted 2023-12-20 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Lung Neoplasms
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Genistein; Paclitaxel; Carboplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single-arm (Experimental): Ascending dose evaluation of BIO 300 Oral Suspension (3 dose levels) given in combination with paclitaxel/carboplatin and radiotherapy.
  Interventions: Drug: BIO 300 Oral Suspension; Drug: Paclitaxel; Drug: Carboplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: BIO 300 Oral Suspension — Cohort 1: BIO 300 500 mg Cohort 2: BIO 300 1,000 mg Cohort 3: BIO 300 1,500 mg Cohort 4: BIO 300 Optimal dose (TBD) BIO 300 dose will be given daily, 7 days/week (Week 1, day 1 through week 6) The 2nd and 3rd dosing cohort (1,000 and 1,500 mg/day) will begin following the accrual of a minimum of 6 subjects at the previous dose level, dose escalation to the next BIO 300 dose level will be allowed to occur when a cohort has completed concurrent chemoradiotherapy with fewer than 33% Dose Limiting Toxicities (DLTs) attributed to BIO 300 Oral Suspension.
  Other Names: genistein, 5, 7-dihydroxy-3-(4-hydroxyphenyl)-chromen-4-one
Drug: Paclitaxel — During the Concurrent Therapy period, paclitaxel 45 mg/m2 will be administered by intravenous drip weekly during weeks 1-6.
  During the Consolidation Therapy period, paclitaxel 200 mg/m2 will be administered by intravenous drip two times, 21 days apart.
  Other Names: Onxol; Taxol
Drug: Carboplatin — During the Concurrent Therapy period, area under the curve (AUC) = 2mg* min/mL will be administered by intravenous drip weekly during weeks 1-6.
  During the Consolidation Therapy period, carboplatin AUC = 6mg*min/mL will be administered by intravenous drip two times, 21 days apart.
  Other Names: Paraplatin; CARBOplatin Novaplus
Radiation: Radiotherapy — Radiation treatment will be scheduled at the discretion of the investigator provided the subject has completed a minimum of 2 days of BIO 300 dosing. Subjects will receive radiation therapy 5 days per week, once daily fractions, 1.8-2.0 Gy per fraction, for 6-7 weeks.

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of BIO 300 Oral Suspension when used in combination with standard dose radiation therapy and chemotherapy in patients with non-small cell lung cancer. Based on preclinical data the investigators hypothesize that BIO 300 Oral Suspension will reduce the incidence of radiation-induced pneumonitis and pulmonary fibrosis.

DETAILED DESCRIPTION:
This is an open-label, single-arm, ascending dose Phase I/II study of BIO 300 Oral Suspension given in combination with paclitaxel/carboplatin and radiotherapy in subjects with stage II, III, or IV NSCLC who are candidates for combined chemoradiotherapy.

A minimum of 6 subjects will be accrued sequentially at each dose level of BIO 300. BIO 300 will be administered daily for the entire course of concurrent chemoradiotherapy, a minimum of 6 weeks; in combination with standard paclitaxel / carboplatin chemotherapy and radiotherapy.

The initial dose of BIO 300 will be administered on Day 1, Visit 2 in which safety data (adverse events, electrocardiograms (ECGs), results of safety laboratory determinations), pharmacokinetic (PK) and pharmacodynamic (PD) data will be collected. PK data will be collected from a minimum of six (6) study subjects from each cohort. PD data will be collected from all subjects in each study cohort. Day 1 of chemotherapy will be scheduled at the discretion of the investigator provided the subject has completed a minimum of 1 day of BIO 300 dosing. BIO 300 will be administered in combination with the chemotherapy components of the protocol (paclitaxel and carboplatin). During the first or second chemotherapy infusion, additional safety, PK and PD data will be collected. Day 1 of radiation therapy (RT) may be scheduled at the discretion of the investigator provided the subject has completed a minimum of 2 days of BIO 300 dosing. BIO 300 will continue to be administered daily; paclitaxel and carboplatin will be administered weekly and radiotherapy will be administered daily until a total dose of 60-70 Gy has been administered. During the period of combined BIO 300 and chemoradiotherapy (6-7 weeks), additional safety, PK and PD data will be collected weekly. An interim data analysis will be completed once the highest dose cohort concludes chemoradiation therapy, in an effort to determine the optimal biological dose. Following analysis, there will be an option to enroll up to an additional 12 subjects at the optimal biological dose. At the conclusion of the study, primary and secondary outcome measures will be evaluated. Data will be analyzed from all cohorts to determine the oncologic response, safety of BIO 300, and a recommended BIO 300 dose.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological confirmation of NSCLC
2. Stage II, III, or IV NSCLC for whom radiation therapy of 60 Gy and concurrent weekly paclitaxel/carboplatin is recommended
3. Up to three small (≤ 3 cm each) lung oligometastases will be allowed and/or one oligometastasis at any other site in the body
4. Eastern Cooperative Oncology Group Performance Scale (ECOG PS) of 0 or 1
5. Forced expiratory volume at one second (FEV1): best value obtained pre- or post-bronchodilator must be ≥ 1.0 liters/second or > 50% predicted value
6. Adequate bone marrow reserve
7. Adequate hepatic reserve
8. Adequate renal function
9. Female subjects of childbearing potential must have a negative pregnancy test
10. Female subjects of childbearing potential and male subjects with female sexual partners of childbearing potential must agree to use an effective method of contraception
11. Ability to read and provide written informed consent

Exclusion Criteria:

1. Weight loss greater than 10% in prior 4 weeks
2. Prior malignancy in which they received any thoracic radiotherapy unless the treating physician considers it unlikely to impact the clinical outcome of the patient
3. Patients with concurrent invasive malignancy other than non-melanoma skin cancer or cervical intraepithelial neoplasia unless the treating physician considers it unlikely to impact the clinical outcome of the patient
4. An active infection or with a fever ≥ 38.5°C
5. Poorly controlled intercurrent illnesses
6. Patients with a prior thoracotomy within 1 week of study registration
7. Chronic Obstructive Pulmonary Disease (COPD) exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days before registration
8. Patients with any of the following are not eligible:

   * Previous history of Corrected QT Interval (QTc ) prolongation resulting from medication that required discontinuation of that medication
   * Congenital long QT syndrome, or 1st degree relative with unexplained sudden death under 40 years of age;
   * Presence of left bundle branch block (LBBB);
   * QTc with Fridericia's correction that is unmeasurable, or ≥ 480 msec on screening ECG. The average QTc from the screening ECG (completed in triplicate) must be < 480 msec in order for the patient to be eligible for the study;
   * Subjects taking any concomitant medication that may cause QTc prolongation, induce Torsades de Pointes are not eligible if QTc ≥ 460 msec.
9. Patients must not have had a clinically significant cardiac event within 6 months before entry; or the presence of any other uncontrolled cardiovascular conditions that, in the opinion of the Investigator, increases the risk of ventricular arrhythmia.
10. Patients with a history of arrhythmia or asymptomatic sustained ventricular tachycardia are not eligible. Patients with atrial fibrillation with well-controlled ventricular rate on medication, are eligible.
11. Psychiatric conditions, social situations or substance abuse that precludes the ability of the subject to cooperate with the requirements of the trial and protocol therapy
12. Grade 2 or higher peripheral neuropathy
13. Known history of Human Immunodeficiency Virus/Acquired Immune Deficiency Syndrome (HIV/AIDS), hepatitis B or C.
14. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception
15. Women who are breastfeeding are not eligible for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-11; Primary Completion 2019-04 (Actual); Study Completion 2020-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D. Kaytor, PhD, Study Director — Humanetics Corporation
Locations (4):
- United States (4):
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Zablocki VA Medical Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simone CB 2nd, Serebrenik AA, Gore EM, Mohindra P, Brown SL, Wang D, Chetty IJ, Vujaskovic Z, Menon S, Thompson J, Fine G, Kaytor MD, Movsas B. Multicenter Phase 1b/2a Clinical Trial of Radioprotectant BIO 300 Oral Suspension for Patients With Non-Small Cell Lung Cancer Receiving Concurrent Chemoradiotherapy. Int J Radiat Oncol Biol Phys. 2024 Feb 1;118(2):404-414. doi: 10.1016/j.ijrobp.2023.08.048. Epub 2023 Aug 29. PMID 37652301
- [Derived] Citrin DE, Prasanna PGS, Walker AJ, Freeman ML, Eke I, Barcellos-Hoff MH, Arankalayil MJ, Cohen EP, Wilkins RC, Ahmed MM, Anscher MS, Movsas B, Buchsbaum JC, Mendonca MS, Wynn TA, Coleman CN. Radiation-Induced Fibrosis: Mechanisms and Opportunities to Mitigate. Report of an NCI Workshop, September 19, 2016. Radiat Res. 2017 Jul;188(1):1-20. doi: 10.1667/RR14784.1. Epub 2017 May 10. PMID 28489488

RESULTS

PARTICIPANT FLOW:
Groups:
- BIO 300 Oral Suspension (500 mg/Day): BIO 300 Oral Suspension (500 mg/day) was given daily, 7 days/week (Week 1, day 1 through the end of concurrent chemoradiotherapy, Weeks 6-7).
- BIO 300 Oral Suspension (1000 mg/Day): BIO 300 Oral Suspension (1000 mg/day) was given daily, 7 days/week (Week 1, day 1 through the end of concurrent chemoradiotherapy, Weeks 6-7).
- BIO 300 Oral Suspension (1500 mg/Day): BIO 300 Oral Suspension (1500 mg/day) was given daily, 7 days/week (Week 1, day 1 through the end of concurrent chemoradiotherapy, Weeks 6-7).
Period: Concurrent Chemoradiotherapy
Arm/Group | BIO 300 Oral Suspension (500 mg/Day) | BIO 300 Oral Suspension (1000 mg/Day) | BIO 300 Oral Suspension (1500 mg/Day)
Started | 7 | 7 | 7
Completed | 6 | 4 | 6
Not Completed | 1 | 3 | 1
Not completed — Death | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Progressive Disease | 0 | 2 | 1
Period: Follow-up
Arm/Group | BIO 300 Oral Suspension (500 mg/Day) | BIO 300 Oral Suspension (1000 mg/Day) | BIO 300 Oral Suspension (1500 mg/Day)
Started | 6 | 4 | 6
Completed | 4 | 3 | 2
Not Completed | 2 | 1 | 4
Not completed — Death | 1 | 0 | 1
Not completed — Progressive Disease | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BIO 300 Oral Suspension (500 mg/Day) | BIO 300 Oral Suspension (1000 mg/Day) | BIO 300 Oral Suspension (1500 mg/Day) | Total
Number analyzed (Participants) | 7 | 7 | 7 | 21
Age, Continuous [Median (Full Range); unit: years] | 78 [69 to 84] | 69 [57 to 83] | 57 [50 to 76] | 69 [50 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 1 | 11
  Male | 2 | 2 | 6 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 3
  Not Hispanic or Latino | 6 | 5 | 7 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 6 | 7 | 6 | 19
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 7 | 21
Initial Tumor Stage [Count of Participants; unit: Participants] — Tumors were staged using the American Joint Committee on Cancer (AJCC) TNM system. The lower the lung cancer stage, the less the cancer has spread and the better the prognosis.
  Participants
    Stage II | 2 | 2 | 1 | 5
    Stage III | 5 | 5 | 4 | 14
    Stage IV | 0 | 0 | 2 | 2
Tumor Histology [Count of Participants; unit: Participants]
  Squamous | 3 | 3 | 4 | 10
  Adenocarcinoma | 4 | 4 | 3 | 11
Primary Tumor Location [Count of Participants; unit: Participants]
  Left Upper Lobe | 3 | 3 | 1 | 7
  Left Lower Lobe | 0 | 1 | 2 | 3
  Right Upper Lobe | 3 | 2 | 4 | 9
  Right Middle Lobe | 0 | 1 | 0 | 1
  Right Lower Lobe | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With BIO 300 Oral Suspension-related Dose Limiting Toxicity
Description: Adverse events of CTCAE v4.0 grade 3 or higher that were possibly, probably or definitely related to BIO 300 Oral Suspension and have occurred before or during concurrent chemoradiotherapy were considered dose limiting toxicities.
Time Frame: Day 1 up to 6 weeks or maximum tolerated dose
Measure: Count of Participants; unit: Participants
Arm/Group | BIO 300 Oral Suspension (500 mg/Day) | BIO 300 Oral Suspension (1000 mg/Day) | BIO 300 Oral Suspension (1500 mg/Day)
Number analyzed (Participants) | 6 | 7 | 7
Participants
  Number of Participants Experiencing DLTs | 0 | 0 | 0
  Number of Participants That Did Not Experience a DLT | 6 | 7 | 7

2. Secondary Outcome: Number of Participants With Adverse Events Throughout the Study
Time Frame: Day 1 up to month 13 post radiation or 12 months post chemotherapy consolidation for surgical participants.
Measure: Number; unit: Participants
Arm/Group | BIO 300 Oral Suspension (500 mg/Day) | BIO 300 Oral Suspension (1000 mg/Day) | BIO 300 Oral Suspension (1500 mg/Day)
Number analyzed (Participants) | 7 | 7 | 7
Participants | 7 | 7 | 7

3. Secondary Outcome: Mean Maximum Serum Concentration (Cmax) of BIO 300 Administered in the Absence of Chemotherapy
Time Frame: Day 1, prior to 1st dose then 0.5, 1, 2, 3, 4, 8 and 24 hours post dose
Population: Only participants that had blood draws for pharmacokinetics were analyzed
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | BIO 300 Oral Suspension (500 mg/Day) | BIO 300 Oral Suspension (1000 mg/Day) | BIO 300 Oral Suspension (1500 mg/Day)
Number analyzed (Participants) | 6 | 6 | 7
ng/mL | 174 (74) | 302 (194) | 388 (264)

4. Secondary Outcome: Mean Area Under the Serum Concentration Curve (AUC) of BIO 300 Administered in the Absence of Chemotherapy
Time Frame: Day 1, prior to 1st dose then 0.5, 1, 2, 3, 4, 8 and 24 hours post dose
Population: Only participants that had blood draws for pharmacokinetics were analyzed
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | BIO 300 Oral Suspension (500 mg/Day) | BIO 300 Oral Suspension (1000 mg/Day) | BIO 300 Oral Suspension (1500 mg/Day)
Number analyzed (Participants) | 6 | 6 | 7
ng*hr/mL | 857 (341) | 1493 (1123) | 1570 (883)

5. Secondary Outcome: Mean Maximum Serum Concentration (Cmax) of BIO 300 When Administered in Combination With Paclitaxel and Carboplatin
Time Frame: Week 1 or 2, during the 1st or 2nd chemotherapy infusion, prior to 1st dose then 0.5, 1, 2, 3, 4, 8, and 24 hours post dose
Population: Only participants that had blood draws for pharmacokinetics were analyzed
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | BIO 300 Oral Suspension (500 mg/Day) | BIO 300 Oral Suspension (1000 mg/Day) | BIO 300 Oral Suspension (1500 mg/Day)
Number analyzed (Participants) | 6 | 6 | 7
ng/mL | 155 (30) | 427 (339) | 414 (257)

6. Secondary Outcome: Mean Area Under the Serum Concentration Curve (AUC) of BIO 300 When Administered in Combination With Paclitaxel and Carboplatin
Time Frame: as for outcome 5
Population: Only participants that had blood draws for pharmacokinetics were analyzed
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | BIO 300 Oral Suspension (500 mg/Day) | BIO 300 Oral Suspension (1000 mg/Day) | BIO 300 Oral Suspension (1500 mg/Day)
Number analyzed (Participants) | 6 | 6 | 7
ng*hr/mL | 1371 (1174) | 1578 (726) | 1821 (964)

7. Secondary Outcome: Mean Maximum Serum Concentration (Cmax) of Paclitaxel When Administered in Combination With BIO 300
Time Frame: Week 1 or 2, during the 1st or 2nd chemotherapy infusion, prior to BIO 300 dose then 0.5, 1, 2, 3, 4, 8 and 24 hours post initial dose
Population: Only participants that had blood draws for pharmacokinetics were analyzed
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | BIO 300 Oral Suspension (500 mg/Day) | BIO 300 Oral Suspension (1000 mg/Day) | BIO 300 Oral Suspension (1500 mg/Day)
Number analyzed (Participants) | 6 | 6 | 3
ng/mL | 665.5 (588.06) | 1026.5 (260.36) | 307.6 (288.2)

8. Secondary Outcome: Mean Area Under the Serum Concentration Curve (AUC) of Paclitaxel When Administered in Combination With BIO 300
Time Frame: as for outcome 7
Population: Only participants that had blood draws for pharmacokinetics were analyzed
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | BIO 300 Oral Suspension (500 mg/Day) | BIO 300 Oral Suspension (1000 mg/Day) | BIO 300 Oral Suspension (1500 mg/Day)
Number analyzed (Participants) | 6 | 6 | 3
ng*hr/mL | 1236.51 (680.63) | 1796.1 (409.49) | 755.27 (306.45)

9. Secondary Outcome: Mean Maximum Serum Concentration (Cmax) of Carboplatin When Administered in Combination With BIO 300
Time Frame: as for outcome 7
Population: Only participants that had blood draws for pharmacokinetics were analyzed
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | BIO 300 Oral Suspension (500 mg/Day) | BIO 300 Oral Suspension (1000 mg/Day) | BIO 300 Oral Suspension (1500 mg/Day)
Number analyzed (Participants) | 6 | 6 | 3
ng/mL | 7594 (1946.03) | 9938.33 (3452.58) | 12883.33 (7446.87)

10. Secondary Outcome: Mean Area Under the Serum Concentration Curve (AUC) of Carboplatin When Administered in Combination With BIO 300
Time Frame: Week1 or 2, during the 1st or 2nd chemotherapy infusion, prior to BIO 300 dose then 0.5, 1, 2, 3, 4, 8 and 24 hours post initial dose
Population: Only participants that had blood draws for pharmacokinetics were analyzed
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | BIO 300 Oral Suspension (500 mg/Day) | BIO 300 Oral Suspension (1000 mg/Day) | BIO 300 Oral Suspension (1500 mg/Day)
Number analyzed (Participants) | 6 | 6 | 3
ng*hr/mL | 30810.04 (5729.8) | 41785.18 (11133.8) | 41753.3 (14462.78)

11. Secondary Outcome: Percent Change From Baseline in Expression Levels of Serum TGF-beta Isoform 1 (TGFB1)
Description: Measuring change from baseline (screening visit) of TGF-beta isoform 1 (TGFB1)
Time Frame: Screening, once weekly during weeks 1-6 of concurrent chemoradiotherapy prior to BIO 300, paclitaxel, and carboplatin dose, and once at the end of consolidation, 3 months and 6 months after the completion of RT
Population: Analysis population only includes subjects that had a baseline measurement during the screening visit
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | BIO 300 Oral Suspension (500 mg/Day) | BIO 300 Oral Suspension (1000 mg/Day) | BIO 300 Oral Suspension (1500 mg/Day)
Number analyzed (Participants) | 6 | 6 | 5
Percent change from baseline
  Week 1: number analyzed (Participants) | 6 | 2 | 5
  Week 1 | 141.8 (64.1) | 96.7 (5.1) | 117.3 (48.5)
  Week 2 | 130.3 (79.9) | 127.5 (77.9) | 96.7 (38.8)
  Week 3 | 108.6 (79.0) | 60.1 (40.1) | 74.4 (25.9)
  Week 4 | 90.6 (66.0) | 69.0 (43.8) | 55.8 (19.9)
  Week 5: number analyzed (Participants) | 6 | 5 | 5
  Week 5 | 88.5 (86.8) | 61.7 (44.3) | 51.2 (12.1)
  Week 6: number analyzed (Participants) | 6 | 2 | 2
  Week 6 | 142.8 (133.9) | 69.3 (43.9) | 33.4 (33.5)
  After consolidation therapy: number analyzed (Participants) | 5 | 4 | 3
  After consolidation therapy | 68.7 (44.2) | 74.3 (78.5) | 60.8 (28.4)
  3 months post-RT: number analyzed (Participants) | 6 | 4 | 3
  3 months post-RT | 205.7 (161.2) | 144.9 (96.4) | 83.1 (18.7)
  6 months post-RT: number analyzed (Participants) | 4 | 2 | 3
  6 months post-RT | 106.5 (57.4) | 130.5 (93.5) | 61.2 (36.6)

12. Secondary Outcome: Rate of Progressive Disease Evaluated by the Response Evaluation Criteria in Solid Tumors (RECIST) (1.1) Criteria
Description: Best Response Rate reported per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by chest CT imaging: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD), At least a 20% increase in the sum of diameters of target lesions; Stable Disease (SD), Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Screening, visits 20, 37, 38, 39, 40, 41 & 42 (through visit 41 for surgical participants)
Measure: Count of Participants; unit: Participants
Arm/Group | BIO 300 Oral Suspension (500 mg/Day) | BIO 300 Oral Suspension (1000 mg/Day) | BIO 300 Oral Suspension (1500 mg/Day)
Number analyzed (Participants) | 6 | 7 | 7
Participants
  Complete Response | 0 | 2 | 2
  Partial Response | 5 | 2 | 2
  Stable Disease | 1 | 3 | 3
  Progressive Disease | 0 | 0 | 0

13. Secondary Outcome: Change in Tumor Diameter as Measured by Diagnostic Computerized Tomography (CT) Scan
Description: Tumor diameter was measured in centimeters. Mean change in tumor diameter from the baseline measurement at screening is reported.
Time Frame: Screening, visits 20 and 3, 6, 11 & 13 months post radiation therapy
Population: Number of participants vary based on the number of subjects that completed a CT scan each timepoint
Measure: Mean (Standard Deviation); unit: Mean Change from Baseline (cm)
Arm/Group | BIO 300 Oral Suspension (500 mg/Day) | BIO 300 Oral Suspension (1000 mg/Day) | BIO 300 Oral Suspension (1500 mg/Day)
Number analyzed (Participants) | 6 | 7 | 7
Mean Change from Baseline (cm)
  Visit 20: number analyzed (Participants) | 6 | 5 | 7
  Visit 20 | -1.30 (1.20) | 0.04 (3.24) | -1.15 (1.63)
  3 Months Post-RT: number analyzed (Participants) | 6 | 5 | 5
  3 Months Post-RT | -2.83 (1.35) | -2.29 (0.82) | -3.54 (1.86)
  6 Months Post-RT: number analyzed (Participants) | 4 | 4 | 5
  6 Months Post-RT | -2.43 (0.99) | -3.23 (1.02) | -3.42 (2.08)
  9 Months Post-RT: number analyzed (Participants) | 4 | 2 | 4
  9 Months Post-RT | -2.58 (0.87) | -3.25 (0.49) | -5.0 (1.75)
  11 Months Post-RT: number analyzed (Participants) | 4 | 3 | 1
  11 Months Post-RT | -2.55 (0.95) | -3.10 (0.56) | -5.9 (0)
  13 Months Post-RT: number analyzed (Participants) | 4 | 3 | 2
  13 Months Post-RT | -2.33 (1.31) | -3.13 (1.27) | -3.05 (5.02)

14. Secondary Outcome: DLCO as Measured by Pulmonary Function Test (PFT)
Time Frame: Screening and months 6 & 13 post radiation therapy completion
Population: Number of participants varies based on the number of study subjects that received each assessment
Measure: Mean (Standard Deviation); unit: mL/mmHg/Min
Arm/Group | BIO 300 Oral Suspension (500 mg/Day) | BIO 300 Oral Suspension (1000 mg/Day) | BIO 300 Oral Suspension (1500 mg/Day)
Number analyzed (Participants) | 7 | 7 | 7
mL/mmHg/Min
  Baseline | 12.12 (3.80) | 14.96 (3.28) | 16.15 (6.60)
  6 months post-RT: number analyzed (Participants) | 4 | 3 | 5
  6 months post-RT | 10.83 (4.31) | 10.46 (4.27) | 11.28 (5.82)
  13 months post-RT: number analyzed (Participants) | 4 | 5 | 2
  13 months post-RT | 11.65 (4.61) | 9.48 (1.92) | 18.95 (1.09)

15. Secondary Outcome: Number of Participants With Pulmonary Fibrosis Assessed by Four-dimensional Computerized Tomography (4D-CT)
Time Frame: Screening, visits 20 & 37 and 9 & 13 months post radiation therapy for non-surgical participants; screening only for surgical participants
Measure: Count of Participants; unit: Participants
Arm/Group | BIO 300 Oral Suspension (500 mg/Day) | BIO 300 Oral Suspension (1000 mg/Day) | BIO 300 Oral Suspension (1500 mg/Day)
Number analyzed (Participants) | 7 | 7 | 7
Participants | 0 | 0 | 0

16. Secondary Outcome: Quality of Life (QOL) as Measured by Functional Assessment of Cancer Therapy-Lung Scale Trial Outcome Index (FACT-L TOI) Patient Reported Outcome Questionnaire.
Description: The Functional Assessment of Cancer Therapy-Lung Scale Trial Outcome Index (FACT-L TOI) questionnaire is a 36-item self-reporting instrument that measures quality of life specific to patients with cancer. Items are rated on a 5 item (point) Likert Scale, from 0 (not at all) to 4 (very much). Total scores range from 0 to 136 and higher scores indicate better quality of life. The FACT-L TOI questionnaire was scored according to FACT-L Scoring Guidelines Version 4.
Time Frame: Screening and months 3, 6, & 13 post radiation therapy completion
Population: Number of participants at each time point vary based on the number of study participants that completed the assessment
Measure: Mean (Standard Deviation); unit: FACT-L Total Score
Arm/Group | BIO 300 Oral Suspension (500 mg/Day) | BIO 300 Oral Suspension (1000 mg/Day) | BIO 300 Oral Suspension (1500 mg/Day)
Number analyzed (Participants) | 7 | 7 | 7
FACT-L Total Score
  Screening | 66.6 (10.8) | 53.8 (21.5) | 53.9 (13.2)
  3 months post-RT: number analyzed (Participants) | 6 | 3 | 5
  3 months post-RT | 54.5 (16.4) | 63.0 (6.7) | 55.6 (13.3)
  6 months post-RT: number analyzed (Participants) | 4 | 3 | 5
  6 months post-RT | 55.4 (15.5) | 49.7 (13.5) | 51.4 (15.0)
  13 months post-RT: number analyzed (Participants) | 4 | 4 | 4
  13 months post-RT | 50.8 (22.4) | 61.5 (18.1) | 55.0 (13.8)

17. Secondary Outcome: Quality of Life (QOL) as Measured by University of California, San Diego-Shortness of Breath Questionnaire (UCSD-SOBQ) Patient Reported Outcome Questionnaire.
Description: The UCSD-SOBQ is a 24-item patient self-reported questionnaire where items are scored on a 6-point scale (0, "not at all" to 5, "maximal or unable to-do because of breathlessness"). Total scores range from 0 to 120 and lower scores indicate better quality of life.
Time Frame: Screening and months 3, 6, & 13 post radiation therapy completion
Population: Number of participants at each time point vary based on the number of study participants that completed the assessment
Measure: Mean (Standard Deviation); unit: UCSD-SOBQ Total Score
Arm/Group | BIO 300 Oral Suspension (500 mg/Day) | BIO 300 Oral Suspension (1000 mg/Day) | BIO 300 Oral Suspension (1500 mg/Day)
Number analyzed (Participants) | 7 | 7 | 7
UCSD-SOBQ Total Score
  Screening | 19.4 (17.4) | 29.9 (32.3) | 13.9 (11.9)
  3 months post-RT: number analyzed (Participants) | 6 | 3 | 5
  3 months post-RT | 37.0 (33.5) | 38.0 (13.9) | 23.0 (20.8)
  6 months post-RT: number analyzed (Participants) | 4 | 3 | 5
  6 months post-RT | 46.8 (31.1) | 54.7 (26.6) | 24.8 (20.8)
  13 months post-RT: number analyzed (Participants) | 4 | 4 | 5
  13 months post-RT | 64.0 (43.6) | 39.8 (23.4) | 23.2 (18.0)

18. Secondary Outcome: Extent of Esophagitis by Patient Reported Swallowing Diary
Description: The assessment will provide a score (the swallowing questionnaire) from 0 to 5; 1 no problems swallowing; 2 mild soreness only; 3 some difficulty swallowing solids; 4 cannot swallow solids; and 5 cannot swallow liquids.
Time Frame: Screening, weeks 1, 2, 3, 4, 5, & 6 and months 3 & 6 post radiation therapy completion
Population: Number of participants at each time point vary based on the number of study participants that completed the assessment
Measure: Mean (Standard Deviation); unit: Swallowing Diary Score
Arm/Group | BIO 300 Oral Suspension (500 mg/Day) | BIO 300 Oral Suspension (1000 mg/Day) | BIO 300 Oral Suspension (1500 mg/Day)
Number analyzed (Participants) | 5 | 7 | 6
Swallowing Diary Score
  Weeks 1-6 Average | 1.2 (0.36) | 1.54 (0.41) | 1.64 (0.87)
  3 months post-RT: number analyzed (Participants) | 5 | 3 | 5
  3 months post-RT | 1.0 (0) | 1.0 (0) | 1.6 (0.89)
  6 months post-RT: number analyzed (Participants) | 3 | 3 | 5
  6 months post-RT | 1.33 (0.58) | 1.0 (0) | 1.6 (0.55)

19. Secondary Outcome: Mean Weekly BIO 300 Trough Levels, Serum Concentration of BIO 300
Time Frame: Concurrent chemoradiotherapy weeks 1, 2, 3, 4, 5 and 6
Population: Number of participants analyzed at each time point varies based on the number of subjects available for pharmacokinetic blood draw
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | BIO 300 Oral Suspension (500 mg/Day) | BIO 300 Oral Suspension (1000 mg/Day) | BIO 300 Oral Suspension (1500 mg/Day)
Number analyzed (Participants) | 5 | 6 | 7
ng/mL
  Week 1: number analyzed (Participants) | 5 | 0 | 6
  Week 1 | 44.2 (90.0) |  | 16.02 (23.7)
  Week 2: number analyzed (Participants) | 5 | 5 | 7
  Week 2 | 32.6 (44.2) | 5.84 (8.8) | 9.96 (13.9)
  Week 3 | 5.1 (4.5) | 5.56 (8.0) | 14.12 (18.6)
  Week 4: number analyzed (Participants) | 5 | 5 | 7
  Week 4 | 8.3 (13.9) | 3.82 (6.0) | 22.66 (44.7)
  Week 5: number analyzed (Participants) | 5 | 5 | 7
  Week 5 | 40.7 (36.2) | 6.71 (11.9) | 23.54 (38.0)
  Week 6: number analyzed (Participants) | 5 | 2 | 4
  Week 6 | 12.4 (15.7) | 24.0 (32.5) | 24.54 (23.8)

20. Secondary Outcome: Weekly Paclitaxel Trough Levels, Plasma Concentration of Paclitaxel and Carboplatin
Description: Serum trough levels of paclitaxel and carboplatin were measured. Carboplatin trough levels were below the limit of quantification at all timepoints and are therefore reported as NA (Not Available).
Time Frame: Concurrent chemoradiotherapy weeks 1, 2, 3, 4, 5 and 6
Population: Number of participants at each time point varies based on the number of participants with blood sample available for analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Paclitaxel: All subjects receiving concurrent paclitaxel chemoradiotherapy
- Carboplatin: All subjects receiving concurrent carboplatin chemoradiotherapy
Arm/Group | Paclitaxel | Carboplatin
Number analyzed (Participants) | 13 | 13
ng/mL
  Week 1: number analyzed (Participants) | 4 | 4
  Week 1 | 1.04 (0.08) | NA (NA) — NA (Not Applicable) because measurement was below the limit of quantification.
  Week 2: number analyzed (Participants) | 12 | 10
  Week 2 | 1.09 (0.19) | NA (NA) — NA (Not Applicable) because measurement was below the limit of quantification.
  Week 3 | 1.53 (0.93) | NA (NA) — NA (Not Applicable) because measurement was below the limit of quantification.
  Week 4: number analyzed (Participants) | 11 | 12
  Week 4 | 1.83 (0.81) | NA (NA) — NA (Not Applicable) because measurement was below the limit of quantification.
  Week 5: number analyzed (Participants) | 12 | 11
  Week 5 | 1.90 (0.96) | NA (NA) — NA (Not Applicable) because measurement was below the limit of quantification.
  Week 6: number analyzed (Participants) | 8 | 10
  Week 6 | 1.92 (1.19) | NA (NA) — NA (Not Applicable) because measurement was below the limit of quantification.

21. Secondary Outcome: FVC as Measured by Pulmonary Function Test (PFT)
Time Frame: Screening and months 6 & 13 post radiation therapy completion
Population: Number of participants varies based on the number of study subjects that received each assessment
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | BIO 300 Oral Suspension (500 mg/Day) | BIO 300 Oral Suspension (1000 mg/Day) | BIO 300 Oral Suspension (1500 mg/Day)
Number analyzed (Participants) | 7 | 7 | 7
Liters
  Baseline | 2.46 (0.46) | 2.79 (0.56) | 3.51 (0.85)
  6 months post-RT: number analyzed (Participants) | 4 | 3 | 5
  6 months post-RT | 2.32 (0.65) | 2.1 (0.60) | 2.93 (0.74)
  13 months post-RT: number analyzed (Participants) | 4 | 5 | 2
  13 months post-RT | 2.32 (0.67) | 2.19 (0.44) | 3.28 (0.27)

22. Secondary Outcome: FEV1 as Measured by Pulmonary Function Test (PFT)
Time Frame: Screening and months 6 & 13 post radiation therapy completion
Population: Number of participants varies based on the number of study subjects that received each assessment
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | BIO 300 Oral Suspension (500 mg/Day) | BIO 300 Oral Suspension (1000 mg/Day) | BIO 300 Oral Suspension (1500 mg/Day)
Number analyzed (Participants) | 7 | 7 | 7
Liters
  Baseline | 1.69 (0.38) | 1.91 (0.59) | 2.39 (0.83)
  6 months post-RT: number analyzed (Participants) | 4 | 3 | 5
  6 months post-RT | 1.71 (0.53) | 1.29 (0.13) | 2.03 (0.60)
  13 months post-RT: number analyzed (Participants) | 4 | 5 | 2
  13 months post-RT | 1.61 (0.55) | 1.26 (0.06) | 2.39 (0.27)

ADVERSE EVENTS:
Time Frame: Day 1 up to month 13 post radiation or 12 months post chemotherapy consolidation for surgical participants.
Description: The CTCAE Version 4.03 was used to grade all AEs. All reported terms and descriptions for AEs were coded using CTCAE Version 4.03.
Arm/Group | BIO 300 Oral Suspension (500 mg/Day) | BIO 300 Oral Suspension (1000 mg/Day) | BIO 300 Oral Suspension (1500 mg/Day)
All-Cause Mortality (participants affected / at risk) | 2/7 | 0/7 | 1/7
Serious Adverse Events (participants affected / at risk) | 3/7 | 1/7 | 2/7
Other Adverse Events (participants affected / at risk) | 7/7 | 7/7 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIO 300 Oral Suspension (500 mg/Day) (N=7) | BIO 300 Oral Suspension (1000 mg/Day) (N=7) | BIO 300 Oral Suspension (1500 mg/Day) (N=7)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic Event (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Lower Respiratory Tract Infection/Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIO 300 Oral Suspension (500 mg/Day) (N=7) | BIO 300 Oral Suspension (1000 mg/Day) (N=7) | BIO 300 Oral Suspension (1500 mg/Day) (N=7)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Edema Limbs (General disorders) | 2 (3) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 3 (3) | 4 (4)
Neutrophil Count Decreased (Investigations) | 3 (3) | 5 (5) | 1 (1)
Platelet Count Decreased (Investigations) | 2 (2) | 5 (5) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 5 (5) | 7 (7)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Infusion Related Reaction (General disorders) | 0 (0) | 0 (0) | 2 (2)
Pain (Non-Cardiac) (General disorders) | 0 (0) | 1 (1) | 1 (1)
Radiation Dermatitis (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 4 (4)
Anemia (Investigations) | 1 (1) | 2 (2) | 2 (2)
Lymphocyte Decreased (Investigations) | 0 (0) | 4 (4) | 3 (3)
Serum Amylase Increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Weight Loss (Investigations) | 0 (0) | 1 (1) | 3 (3)
White Blood Cell Decreased (Investigations) | 1 (1) | 6 (6) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypomagnesemi (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Tremors (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2)
Dry Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 3 (3)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-26): https://cdn.clinicaltrials.gov/large-docs/99/NCT02567799/Prot_SAP_000.pdf